CLINICAL TRIAL: NCT06979219
Title: Streamlining Radioembolization for HCC ≤ 5 cm With Y90 Resin Microspheres : Multicenter Prospective Registry Study
Brief Title: Streamlining Radioembolization for Small HCC
Acronym: ISTAR-02
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Cheol Kim, Clinical Professor, Seoul National University Hospital
Other Study IDs: 2503-052-1620
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Streamlining group: radioembolization is performed without MAA scan

SUMMARY:
In patients who has no sign suggesting high lung shunt fraction (TIPS, hepatic vein invasion, hepatic vein enhancement on arterial phase, dysmorphic intratumoral vessel, tumor size < 5cm), radioembolization is performed without MAA scan with SIR-Spheres. This prospective registry will prove that the selection criteria is accurate and streamlining radioembolization is feasible and safe.

ELIGIBILITY:
Inclusion Criteria:

* HCC can be diagnosed by AASLD guideline
* hepatocellular carcinoma 5cm or smaller
* dysmorphic intratumoral vessels 3mm or smaller
* Child-Pugh class A
* ECOG 0 or 1
* the following lab should be met. A. Leukocytes ≥ 1,000/µL and ≤ 20,000/µL B. Hemoglobin ≥ 6.0 g/dL (transfusion allowed to meet this criterion) C. Total bilirubin ≤ 2.0 mg/dL D. Platelet ≥ 40,000/µL E. International normalized ratio (INR) ≤ 2.0 for patients not taking anticoagulants F. Aspartate transaminase (AST) ≤ 800 IU/L (i.e., ≤ 20X upper normal limit) G. Alanine transaminase (ALT) ≤ 800 IU/L (i.e., ≤ 20X upper normal limit) H. Creatinine ≤ 2.5 mg/dL (if patient is receiving hemodialysis, no upper limit of creatinine)

Exclusion Criteria:

* hepatic vein invasion on CT/MRI
* hepatic vein enhancement on arterial phase of CT/MRI
* TIPS
* dysmorphic intratumoral vessels > 3mm
* main portal vein invasion
* significant COPD or interstitial lung disease
* biliary stent or bilioenteric anastomosis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with hepatocellular carcinoma who are scheduled for radioembolization
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
complete response rate by mRECIST | up to 1 year
  the proportion of CR by mRECIST at any time of the primary target tumor

SECONDARY OUTCOMES:
objective response rate | up to 1 year
local progression-free survival | From date of radioembolization until the date of first documented progression of treated tumor or date of death from any cause, whichever came first, assessed up to 60 months
Progression-free survival | From date of radioembolization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
overall survival | From date of radioembolization until the date of death from any cause, assessed up to 60 months

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - National Cancer Center, Goyang
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance hospital, Seoul

IPD SHARING:
Plan to Share IPD: No